CLINICAL TRIAL: NCT01359722
Title: N-acetylcysteine to Prevent Renal Failure in Patients With Chronic Kidney Disease Undergoing Coronary Artery Bypass Surgery
Brief Title: N-acetylcysteine to Prevent Renal Failure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto do Coracao (Other Government)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: José Jayme Galvão de Lima, Instituto do Coracao
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 0992/09
Record Dates: First submitted 2011-05-18; First posted 2011-05-25 (Estimated); Last update posted 2011-05-25 (Estimated); Status verified 2009-10

CONDITIONS: Kidney Failure, Acute; Oxidative Stress Induction
Keywords: N-acetylcysteine; Myocardial Revascularization; Acute Renal Failure; Oxidative Stress
MeSH Terms: conditions — Acute Kidney Injury | interventions — Acetylcysteine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- N-Acetylcysteine (Experimental): N-acetylcysteine is administered at a dose of 150mg/kg in 500mL of saline EV in 1 hour followed by a dose of 50mg/kg in 500 mL of saline IV within 6 hours, beginning the infusion together to surgery.
  Interventions: Drug: N-acetylcysteine
- Control (Placebo Comparator): This group will receive only the infusion of saline in the same doses and infusion rate.
  Interventions: Drug: Control

INTERVENTIONS:
Drug: N-acetylcysteine — N-acetylcysteine is administered at a dose of 150mg/kg in 500mL of saline EV in 1 hour followed by a dose of 50mg/kg in 500 mL of saline IV within 6 hours, beginning the infusion together to surgery.
  Other Names: Fluimucil
  Arms: N-Acetylcysteine
Drug: Control — The control group will receive only the infusion of saline in the same doses and infusion rate.
  Other Names: saline
  Arms: Control

SUMMARY:
The purpose of this study is to determine the possible effect nephroprotective of N-acetylcysteine in patients with chronic kidney disease undergoing elective coronary artery bypass grafting by serial evaluation of renal function and to evaluate whether treatment reduces cardiac mortality, cardiac events and Global mortality, if it interferes with oxidative stress and inflammation and the need for dialysis.

DETAILED DESCRIPTION:
Renal failure is a serious and relatively frequent complication of cardiac surgery was observed, especially in diabetics and those with pre-existing renal dysfunction. Given that oxidative stress is elevated in diabetics and in renal and heart, it is reasonable to speculate on its involvement in the pathophysiology of this complication. It is unknown whether the incidence of postoperative renal failure can be reduced by antioxidants. N-acetylcysteine (NAC) is an antioxidant that prevents nephropathy induced by contrast medium and aminoglycosides and increases intracellular levels of cyclic guanosine monophosphate, acting as a vasodilator and platelet inhibitor.

Based on a knowledge of the pathophysiology of ARF, several interventions have been attempted over the past decades. However, various measures employed successfully in the prevention of experimental ARF did not result in success in clinical practice. Much of this failure is probably due to the difference between the experimental models of ARF that encountered in the clinic. Other factors that should be considered, and that may explain the poor results in clinical trials are: the time of use of the drug, dosage and route of administration, are not always adequate.

From the data in the literature, it remains doubtful whether the protective role of NAC is limited only to contrast nephropathy or whether it could have application in other clinical situations in which oxidative stress and vasoconstriction are determinants of injury, as occurs, for example, in CABG surgeries.

NAC is a drug of low cost and low toxicity, this paper intend to assess its role as prophylaxis of renal dysfunction in the postoperative period of CABG in patients with chronic kidney disease stages 3 and 4 (GFR between 15 and 59 mL/min/1, 73 m2 of body surface).

ELIGIBILITY:
Inclusion Criteria:

* adult patients aged 30 to 80 years old of both sexes
* indicated for elective CABG
* with glomerular filtration rate, assessed with the MDRD <60 mL/min/1, 73 m2 and> 15 mL / min / 1.73 m2 body surface

Exclusion Criteria:

* patients on chronic dialysis or with creatinine> 5 mg / dL preoperatively; individuals allergic or intolerant to N-acetylcysteine
* pregnant women
* patients with cancer
* patients underwent re-surgery within the first 72 hours postoperatively

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2010-03; Primary Completion 2011-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Decrease in glomerular filtration defined by at least 30% compared to preoperative levels . | Within the first 72 hours postoperatively

SECONDARY OUTCOMES:
Up 50% of preoperative levels of serum creatinine. | Within the first 72 hours after surgery and cardiovascular morbidity and all-cause mortality at thirty days post-operatively.
Death from any cause. | Within the first 72 hours after surgery and cardiovascular morbidity and all-cause mortality at thirty days post-operatively.
Need for dialysis | Within the first 72 hours after surgery and cardiovascular morbidity and all-cause mortality at thirty days post-operatively.
Cardiovascular morbidity. | Within the first 72 hours after surgery and cardiovascular morbidity and all-cause mortality at thirty days post-operatively.
Increased levels of Cystatin C. | Within the first 72 hours after surgery and cardiovascular morbidity and all-cause mortality at thirty days post-operatively.
Increased levels of NGAL. | Within the first 72 hours after surgery and cardiovascular morbidity and all-cause mortality at thirty days post-operatively.
Increased levels of isoprostane. | Within the first 72 hours after surgery and cardiovascular morbidity and all-cause mortality at thirty days post-operatively.

CONTACTS AND LOCATIONS:
Overall Officials: Jose Jayme G de Lima, phD, Principal Investigator — Instito do Coracao-HCFMUSP
Locations (1):
- Instituto do Coracao, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Suen WS, Mok CK, Chiu SW, Cheung KL, Lee WT, Cheung D, Das SR, He GW. Risk factors for development of acute renal failure (ARF) requiring dialysis in patients undergoing cardiac surgery. Angiology. 1998 Oct;49(10):789-800. doi: 10.1177/000331979804900902. PMID 9783643
- [Background] Tepel M, van der Giet M, Schwarzfeld C, Laufer U, Liermann D, Zidek W. Prevention of radiographic-contrast-agent-induced reductions in renal function by acetylcysteine. N Engl J Med. 2000 Jul 20;343(3):180-4. doi: 10.1056/NEJM200007203430304. PMID 10900277
- [Background] Shyu KG, Cheng JJ, Kuan P. Acetylcysteine protects against acute renal damage in patients with abnormal renal function undergoing a coronary procedure. J Am Coll Cardiol. 2002 Oct 16;40(8):1383-8. doi: 10.1016/s0735-1097(02)02308-2. PMID 12392825
- [Background] Mazzon E, Britti D, De Sarro A, Caputi AP, Cuzzocrea S. Effect of N-acetylcysteine on gentamicin-mediated nephropathy in rats. Eur J Pharmacol. 2001 Jul 13;424(1):75-83. doi: 10.1016/s0014-2999(01)01130-x. PMID 11470263
- [Background] Baker CS, Wragg A, Kumar S, De Palma R, Baker LR, Knight CJ. A rapid protocol for the prevention of contrast-induced renal dysfunction: the RAPPID study. J Am Coll Cardiol. 2003 Jun 18;41(12):2114-8. doi: 10.1016/s0735-1097(03)00487-x. PMID 12821233